CLINICAL TRIAL: NCT04428684
Title: COMPARISON OF A NEW FORMULATION OF GOSERELIN (Pepti 3.6 mg) to Zoladex® 3.6 mg IN PATIENTS WITH DYSFUNCTIONAL UTERINE BLEEDING REQUIRING ENDOMETRIAL ABLATION.
Brief Title: COMPARISON OF A NEW FORMULATION OF GOSERELIN (Pepti 3.6 mg) to Zoladex® 3.6 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peptigroupe Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pepti 3.6 E 01
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Dysfunctional Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Goserelin

STUDY DESIGN:
Intervention Model Description: Comparative parallel design aimed at showing non-inferiority
Who Masked: Outcomes Assessor
Masking Description: Sponsor, independant statistician, radiologists and bioanalytical lab are all blinded to treatment regimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pepti 3.6 treatment (Experimental): Patients treated with goserelin depot 3.6 mg. One injection on Day 0 and a second injection on Day 28
  Interventions: Drug: Pepti 3.6 mg
- Zoladex 3.6 mg treatment (Active Comparator): Patients treated with goserelin depot 3.6 mg. One injection on Day 0 and a second injection on Day 28
  Interventions: Drug: Pepti 3.6 mg

INTERVENTIONS:
Drug: Pepti 3.6 mg — Each patient receives one injection of Pepti 3.6mg or Zoladex 3.6mg on Day 0 and a second injection of the same drug given the first time on Day 28. On Day 42 patients undergo endometrial ablation
  Other Names: Zoladex 3.6 mg

SUMMARY:
The comparator drug (Zoladex 3.6 mg) is approved for use as a thinning agent for the endometrium prior to endometrial ablation. The dosing recommendation is one or two depots with each depot given four weeks apart. When two depots are administered, surgery should be performed within two to four weeks following administration of the second depot.

DETAILED DESCRIPTION:
The primary objective of the study is to demonstrate non-inferiority of a generic formulation of goserelin 3.6 mg as compared to Zoladex ® 3.6 mg on endometrial thinning prior to surgery. The study is an open label, multicenter, prospective, parallel group randomized study.

Blind for Sponsor, ultrasound assessment, testing labs and statistician, the study will be performed in premenopausal women with dysfunctional uterine bleeding (DUB) eligible for endometrial ablation. Patients will be randomized in a 1 to 1 ratio to receive either the Peptigroupe test product (Pepti 3.6 mg) or Zoladex® 3.6 mg for a treatment of 8 weeks (two injections).

Ultrasonic measurement of endometrial thickness will be performed on screening and on days 0 (pre-injection), 28 (pre-injection) and 42 (pre surgical procedure).

The pharmacodynamics profile will be tabulated at the end of the study on the basis of the following data:

1. Estradiol
2. LH and FSH as additional information on hormone response

Goserelin safety profile will be assessed throughout the study on the basis of the following assessments:

1. Treatment-emergent AEs
2. Physical examinations
3. Vital signs
4. 12-Lead ECG
5. Laboratory parameters (i.e., biochemistry, haematology, and urinalysis)

ELIGIBILITY:
Inclusion Criteria:

1. Be pre-Menopausal females with regular menstrual cycles and > 30 years of age 2. Premenopausal at enrollment as determined by FSH measurement ≤ 60 IU/mL. 3. Endometrial thickness at pre-treatment less than 20 mm. 4. Diagnosis of Dysfunctional Uterine Bleeding and requiring endometrial ablation 5. Tumour negative cytology and histology 6. Appropriate sized uterus with no anatomic pathologies 7. Patient is not pregnant and does not wish to become pregnant in the future 8. Patient is willing to use a non-hormonal contraception method during the study, nor an intra-uterine device 9. Patient has no endocrine disorders, is not receiving hormonal therapies or non-steroidal anti-inflammatory medication. (prophylactic antibiotics can be administered according to the usual practice of the investigator) 10. Have the ability to understand the requirements of the study and is willing to provide written informed consent 11. Agree to abide by the study restrictions and return for the required assessments 12. Only patients which can be discontinued safely from contra-indicated medications discussed below in section 7.4 can be included in the study.

-

Exclusion Criteria:

1. Be pregnant or have desire to conceive
2. Have abnormal endometrial cytology as confirmed by histology
3. Have active endometritis
4. Have active pelvic inflammatory disease
5. Have active sexually transmitted disease (STD), at the time of ablation. Note: Treatment of STD documented in the chart serves as sufficient evidence of infection resolution. Patient may be considered for study enrollment.
6. Presence of bacteremia, sepsis, or other active systemic infection
7. Have active infection of the genitals, vagina, cervix, uterus or urinary tract at the time of inclusion
8. Known/suspected gynecological malignancy within the past 5 years
9. Known clotting defects or bleeding disorders
10. Untreated/unevaluated cervical dysplasia
11. Known/suspected abdominal/pelvic cancer
12. Atypical Hyperplasia
13. Prior uterine surgery (except low segment cesarean section) that interrupts the integrity of the uterine wall (e.g., myomectomy or classical cesarean section
14. Currently on medications that could thin the myometrial muscle, such as long-term steroid use (except inhaler or nasal therapy for asthma)
15. Currently on anticoagulants
16. Have a known hypersensitivity to gonadotropin releasing hormone (GnRH), GnRH agonists, any LHRH agonists (e.g., leuprolide (Lupron®), goserelin ( Zoladex®) etc.) or to the PLGA polymers contained in the study formulation
17. Have a severe liver disease (e.g., cirrhosis, chronic active hepatitis or chronic persistent hepatitis) or has persistent ALT, AST ˃ 2 X ULN, serum creatinine ˃ 2 X ULN, serum bilirubin ˃ 2 X ULN
18. Have received an investigational drug or participated in a clinical trial within the last 30 days
19. Have clinically serious and/or unstable concurrent infection, medical illnesses or conditions that are uncontrolled or whose control, in the opinion of the Investigator, may be jeopardized by participation in this study or by the complications of this therapy
20. Patients with BMI ˂ 18
21. Anticoagulated patients with INR ≥ 2
22. Patients with a history of QT prolongation, congenital long QT syndrome, electrolyte abnormalities, CHF, or concurrent administration with QT prolonging drugs or QTc ˃450 msec.

    -

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Non-inferiority in terms of activity of test drug versus comparator | 1 year
  Non-inferiority of test drug compared to comparator in terms of reduction of the endometrial thickness prior to surgical ablation

CONTACTS AND LOCATIONS:
Overall Officials: Bonabes deRougé, MD, Study Director — Peptigroupe Inc.; Andrii Zaremba, Study Chair — Pharmaxi LLC
Locations (5):
- Ukraine (5):
  - Central Military Hospital, Kyiv
  - LLC Medical Center, Kyiv
  - Maternity Hospital no 3, Kyiv
  - Center for Innovative Medical Technologies of the National Academy of Sciences, Kyiv
  - City Clinical Hospital, Kyiv

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers